CLINICAL TRIAL: NCT03802812
Title: Thin Bronchoscope and Virtual Bronchoscopic Navigation System for Rapid Detection of Mycobacterium Tuberculosis and Resistant-conferring Mutations
Brief Title: Thin Bronchoscope and Virtual Bronchoscopic Navigation System for Tuberculosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Jeongha Mok, Clinical Professor, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TBVBN study; 2018R1C1B5085364 (Other Grant/Funding Number: National Research Foundation of Korea)
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional arm (No Intervention): Perform bronchial washing using conventional methods.
  * CT-guided thick bronchoscope
- Investigational arm (Active Comparator): Perform bronchial washing using investigational methods.
  * virtual bronchoscopic navigation (VBN)-guided thin bronchoscope (4.0mm of outer diameter)
  Interventions: Device: Thin bronchoscope and VBN

INTERVENTIONS:
Device: Thin bronchoscope and VBN — targeted washing at more adjacent TB lesion using thin bronchoscope and virtual bronchoscopic navigation system
  Arms: Investigational arm

SUMMARY:
This study investigates the utility of thin bronchoscope and virtual bronchoscopic navigation system (targeted bronchial washing) for detection of M. tuberculosis and resistant-conferring mutations in patients with pulmonary tuberculosis. Time to appropriate treatment and stain/culture conversion are also evaluated.

DETAILED DESCRIPTION:
Comparisons of detection rate of M. tuberculosis and resistant-conferring mutations between patients who perform CT-guided conventional bronchoscope and patients who perform VBN-guided thin bronchoscope.

ELIGIBILITY:
Inclusion Criteria:

* age of 18 or more
* persons who are suspected with pulmonary tuberculosis on radiologic examination
* persons who cannot spit sputum or persons with negative results on sputum AFB smear and TB-PCR or Xpert MTB/RIF assay

Exclusion Criteria:

* persons who do not agree with bronchoscopy (persons who want empirical treatment for TB)
* persons with contraindications for bronchoscopy

  * bleeding tendency
  * uncontrolled respiratory disease (hypoxemia)
  * uncontrolled cardiovascular disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
detection of M. tuberculosis and resistant-conferring mutations | 2months after procedure
  evaulation by sensitivity, specificity, PPV and NPV

SECONDARY OUTCOMES:
time to appropriate treatment and stain/culture conversion | 6months after procedure
  date of treatment initiation and stain/culture negative conversion

CONTACTS AND LOCATIONS:
Overall Officials: Jeongha Mok, MD, PhD, Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan National University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eom JS, Park S, Jang H, Kim S, Yoo WH, Kim SH, Mok J. Bronchial Washing Using a Thin Versus a Thick Bronchoscope to Diagnose Pulmonary Tuberculosis: A Randomized Trial. Clin Infect Dis. 2023 Jan 13;76(2):238-244. doi: 10.1093/cid/ciac789. PMID 36151949